CLINICAL TRIAL: NCT04355455
Title: Effects of Serotonin Agonist Citalopram on Multimodal Esophageal Stimulation in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: Citalopram MuMoS HV
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram (Active Comparator): Administration of citalopram to assess the esophageal sensitivity in HV
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Administration of placebo to assess the esophageal sensitivity in HV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — 40 mg citalopram intravenously
  Arms: Citalopram
Drug: Placebo — Saline solution
  Arms: Placebo

SUMMARY:
To investigate the effect of citalopram, a selective serotonin reuptake inhibitor, on esophageal sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* HV aged between 18 - 60 years

Exclusion Criteria:

* history of psychiatric disease or a positive first degree psychiatric family history
* pregnancy or lactation
* concomitant administration of any centrally activating medication (anti-depressive medication, hypnotics, sedatives, anxiolytics, …)
* medication affecting esophageal motility
* significant co-morbidities (neuromuscular, psychiatric, cardiovascular, pulmonary, endocrine, autoimmune, renal and hepatic)
* prior history of esophageal, gastric surgery or endoscopic anti-reflux procedure
* history of gastrointestinal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in sensitivity to thermal stimulation | After 1 hour 30 minutes after administration citalopram, we will start with the thermal stimulation
  To detect changes in thermal stimulation for sensitivity

SECONDARY OUTCOMES:
Change in sensitivity to mechanical stimulation | After 1 hour 45 minutes after administration citalopram, we will start with the mechanical stimulation
  To detect changes in mechanical stimulation for sensitivity
Change in sensitivity to electrical stimulation | After 2 hours after administration citalopram, we will start with the electrical stimulation
  To detect changes in electrical stimulation for sensitivity
Change in sensitivity to chemical stimulation | After 2 hours 15 minutes after administration citalopram, we will start with the chemical stimulation
  To detect changes in chemical stimulation for sensitivity
Change in positive and negative affect score | At the beginning of the study and at the end of the multimodal stimulation
  To detect change in affect of the multimodal stimulation using the PANAS = Positive and Negative Affect scale that consists of two 10-item scales to measure both positive and negative affect. Higher score on the Positive scale is better; Higher score on the Negative Affect scale is worse.
Change in state trait and anxiety score | At the beginning of the study and at the end of the multimodal stimulation
  to detect changes in the score due to the multimodal stimulation using the The State-Trait Anxiety Inventory (STAI). Each type of anxiety has its own scale of 20 different questions that are scored.Scores range from 20 to 80, with higher scores correlating with greater anxiety.

IPD SHARING:
Plan to Share IPD: No